CLINICAL TRIAL: NCT02773199
Title: Effects of Preoperative Fasting on ECG and Vital Parameters in Patients Undergoing Orthopedic and Urologic Surgery
Brief Title: Effects of Preoperative Fasting on ECG and Vital Parameters
Status: Completed | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IzmirBozyaka
Record Dates: First submitted 2016-05-11; First posted 2016-05-16 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Fasting; Intraoperative Complications; Ischemia
MeSH Terms: conditions — Fasting; Intraoperative Complications; Ischemia | interventions — Anesthesia, Spinal; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1- Morning Surgery: Patients' who are scheduled for surgery under spinal anesthesia with bupivacaine in morning hours (until 12pm) will be included in this cohort. Since all patients are ordered to stop oral ingestion by 12am at the day of the surgery, patients in this cohort will be exposed to a preoperative fasting for 8 hours
  Interventions: Other: Preoperative Fasting for 8 hours; Drug: Spinal Anesthesia with Bupivacaine
- Cohort 2- Afternoon Surgery: Patients' who are scheduled for surgery under spinal anesthesia with bupivacaine in afternoon hours (after 12pm) will be included in this cohort. Since all patients are ordered to stop oral ingestion by 12am at the day of the surgery, patients in this cohort will be exposed to a preoperative fasting for more than 12 hours
  Interventions: Other: Preoperative Fasting for more than 12 hours; Drug: Spinal Anesthesia with Bupivacaine

INTERVENTIONS:
Other: Preoperative Fasting for 8 hours — Patients will be exposed to preoperative fasting
  Other Names: Shorter Fasting
  Groups: Cohort 1- Morning Surgery
Other: Preoperative Fasting for more than 12 hours — Patients will be exposed to preoperative fasting
  Other Names: Longer Fasting
  Groups: Cohort 2- Afternoon Surgery
Drug: Spinal Anesthesia with Bupivacaine — Spinal Anesthesia with heavy bupivacaine 0.5% is provided.
  Other Names: Spinal Block

SUMMARY:
This study compares differences in hemodynamic ve ECG parameters of patients undergoing urological or orthopedic surgery under spinal anesthesia. First group will comprise of patients undergoing surgery in the morning hours; thus with a standard fasting duration (8 hours), and the second group will comprise of patients undergoing surgery afternoon; thus having a prolonged fasting duration (>12 hours).

DETAILED DESCRIPTION:
Patients who are scheduled for surgery in surgical wards are routinely fasted after 12am on the day of the surgery regardless of the planned hour of the surgery. This results in a near standard fasting for patients with a planned surgery time in morning hours of the day. However, patients with a planned surgery time in the afternoon hours of the day are fasted more than 12 hours. This situation may not look very important for a healthy young adult but considering that the patient population in a hospital is mostly consisted of sick and elderly people, fasting and associated dehydration may have serious deleterious effects. Our objective is to observe and define these potential deleterious effects with a special focus on cardiovascular system of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 60 years of age
* Patients with an ASA (American Society of Anesthesiologists) physical status score of 1, 2 or 3
* Patients scheduled for elective orthopedic or urological surgery under spinal anesthesia

Exclusion Criteria:

* Patients requiring emergency surgery
* Patients under 60 years of age
* Rejecting to participate in the study
* Contraindications to spinal anesthesia
* Evidence of myocardial ischemia in baseline electrocardiogram prior to surgery
* Conditions mimicking electrocardiographic signs of myocardial ischemia (e.g. electrolyte imbalances such as hypokalemia)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 60 who scheduled for urological or orthopedic surgery under spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Evidence of ischemic changes in 12 lead electrocardiogram | Immediately after, 1, 2, 5 and 15 minutes after injection of bupivacaine for spinal block
  Changes in ST and T waves compared to a baseline preoperative ECG will be monitored and recorded right after spinal block is placed, and at 1st, 2nd, 5th and 15th minutes after spinal injection

SECONDARY OUTCOMES:
Evidence of hypotension confirmed by non-invasive blood pressure measurement | Immediately after, 1, 2, 5 and 15 minutes after injection of bupivacaine for spinal block
  Changes in mean arterial blood pressure will be monitored and a decrease of 10% from baseline mean arterial blood pressure will be recorded as hypotension right after, 1, 2, 5 and 15 minutes after injection of bupivacaine for spinal block spinal block is placed
Evidence of hypertension confirmed by non-invasive blood pressure measurement | Immediately after, 1, 2, 5 and 15 minutes after injection of bupivacaine for spinal block
  Changes in mean arterial blood pressure will be monitored and an increase of 10% from baseline mean arterial blood pressure will be recorded as hypertension right after, 1, 2, 5 and 15 minutes after injection of bupivacaine for spinal block
Evidence of hypoxia confirmed by peripheral oxygen saturation probe | Immediately after, 1, 2, 5 and 15 minutes after injection of bupivacaine for spinal block
  Peripheral oxygen saturation will be continuously monitored and any value less than 90% will be recorded right after spinal block is placed, at first, second, fifth minutes and at 15th minute
Evidence of tachycardia in 12 lead electrocardiogram | Immediately after, 1, 2, 5 and 15 minutes after injection of bupivacaine for spinal block
  A heart rate equal to / higher than 100 will be recorded right after spinal block is placed, at first, second, fifth minutes and again at 15th minute
Evidence of bradycardia in 12-lead electrocardiogram | Immediately after, 1, 2, 5 and 15 minutes after injection of bupivacaine for spinal block
  A heart rate equal to / less than 50 will be recorded right after spinal block is placed, at first, second, fifth minutes and again at 15th minute

CONTACTS AND LOCATIONS:
Overall Officials: Oguzhan Yeniay, MD, Principal Investigator — Izmir Bozyaka Training and Research Hospital
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No